CLINICAL TRIAL: NCT04233281
Title: Kori-tofu Proteins and Blood Glucose Response
Acronym: KoPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Asahimatsu Support BV (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL71213.081.19
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Glucose Intolerance
Keywords: Kori tofu; Glucose response; Pre-diabetics
MeSH Terms: conditions — Glucose Intolerance | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kori-tofu added to a carbohydrate rich meal (Experimental): Kori tofu as part of a carbohydrate rich meal
  Interventions: Other: Kori tofu
- Whey protein added to a carbohydrate rich meal (Active Comparator): Whey protein as part of a carbohydrate rich meal
  Interventions: Other: Whey protein

INTERVENTIONS:
Other: Kori tofu — 16.5 gram Kori-tofu mixed in a high carbohydrate test meal
  Arms: Kori-tofu added to a carbohydrate rich meal
Other: Whey protein — high carbohydrate test meal with whey protein, matched in macronutrient content
  Arms: Whey protein added to a carbohydrate rich meal

SUMMARY:
The study is a randomized, cross-over, double blind, controlled trial in which study participants will visit the research facility on two occasions under fasting conditions with a minimum of 1 week between visits. During each visit, participants will receive a carbohydrate rich test-meal with Kori-tofu (protein) or whey protein. The two meals will be given in randomized order and blood will be collected via a catheter before and up to 3 hours after consumption of the test-meal. Study participants will also wear continuous glucose meters during the trial. They will receive a standardized evening meal prior to each study day and are asked not to drink alcohol or perform heavy exercise the day before. After each test day participants are offered a meal.

DETAILED DESCRIPTION:
There are several types of tofu, an example of a specific type of tofu is called Kori-tofu. Kori-tofu literally means frozen tofu. The production process of Kori-tofu leads to the formation of a higher high molecular weight fraction (HMF) content of the soy proteins. Several clinical studies describe the effects of Kofi-tofu on health. In this study, the aim is to investigate whether Kori-tofu protein affects postprandial blood glucose concentrations in participants with an impaired glucose tolerance.

The primary objective is to investigate whether Kori-tofu protein affects postprandial blood glucose concentrations, when administered as a part of an ordinary high carbohydrate meal. The secondary objective is to investigate whether Kori-tofu protein affects postprandial insulin concentrations.

The study is a randomized, cross-over, double blind, controlled trial in which study participants will visit the research facility on two occasions under fasting conditions. Subjects will receive two different carbohydrate-rich meals, either with added Kori-tofu or whey protein, with a washout period of one week. Blood will be collected via a catheter before and up-to 3 hours after consumption of the test-meal.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 kg/m2
* Having veins suitable for blood sampling via a catheter
* Having one or more of the following criteria:

  * HbA1c> 6%
  * fasting glucose >6.1mmol/L
  * two-hour glucose levels >7.8 mmol/L on the 75-g oral glucose tolerance test.

Exclusion Criteria:

* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery
* Kidney dysfunction (self-reported)
* Use of medication/supplements that may influence the study results, such as med-icines known to interfere with glucose homeostasis (judged by our study doctor)
* Anaemia (Hb values <7.5 for women and <8.5 for men)
* Reported slimming, medically prescribed or other extreme diets
* Reported weight loss or weight gain of > 5 kg in the month prior to pre-study screening
* Not willing to give up blood donation during the study
* Current smokers
* Alcohol intake ≥4 glasses of alcoholic beverages per day
* Abuse of illicit drugs
* Food allergies for products that we use in the study
* Participation in another clinical trial at the same time
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
change in blood glucose levels after a carbohydrate rich meal | blood samples will be taken before and up to 3 hours after test meal consumption
  postprandial test, determine glucose levels in blood samples collected before and after the test meal

SECONDARY OUTCOMES:
change in blood insulin levels after a carbohydrate rich meal | blood samples will be taken before and up to 3 hours after teast meal consumption
  postprandial test, determine insulin levels in blood samples collected before and after the test meal
change in postprandial glucose concentrations after food intake | 1.5 week in total to cover both test days and 3-4 days prior to the test day
  measured by a continuous glucose monitoring device

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No